CLINICAL TRIAL: NCT06180733
Title: Neo-adjuvant Pembrolizumab as an Alternative Treatment for MMRd Uterine Cancer, a Phase II Efficacy Study
Brief Title: Neo-adjuvant Pembrolizumab as an Alternative Treatment for MMRd Uterine Cancer
Acronym: PAM-II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hans W. Nijman, MD PHD, Head of Obstetrics and Gynecology, Prinicpal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAM-UMCG-002; 2022-003922-27 (EudraCT Number)
Record Dates: First submitted 2023-12-04; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Uterine Cancer; MMRd; Grade 3; Clear Cell; Neo-adjuvant; Pembrolizumab
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Lymphoma, Follicular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Primary MMRd endometrial cancer patients (Experimental)
  Interventions: Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab (Keytruda), 200mg IV Q3W for a total of 9 administrations per patient, prior to standard-of-care surgery. Patients will be monitored for response and possible progression using MRI and pipelle biopsies.

SUMMARY:
The goal of this clinical trial is to establish the fraction of patients that achieve a major pathological response (MPR) after 9 cycles of pembrolizumab, with the ultimate aim of informing a follow-up randomized trial.

Participants will receive 9 cycles of pembrolizumab before their standard of care hysterectomy.

DETAILED DESCRIPTION:
Objective: Based on the success of the pilot feasibility study, we propose a phase 2 trial to establish the fraction of patients that achieve a major pathologic response (MPR) after 9 cycles of pembrolizumab, with the ultimate aim of informing a follow-up randomized trial. MPR was chosen as primary endpoint to align with ongoing randomized phase 3 ICB trials on neo-adjuvant vs. adjuvant treatment in other tumor types (e.g. the NADINA trial in melanoma; NCT04949113).

Study design: Patients will be treated with neo-adjuvant pembrolizumab (200mg IV Q3W, for a total of 9 administrations), followed by SoC surgery and adjuvant therapy where indicated. Tumor responses to pembrolizumab will be assessed by a pathologist (primary endpoint) using material from the SoC surgery. In addition, tumor response will be evaluated by MRI (secondary endpoint) after the second, fourth, sixth, and last cycle of pembrolizumab. In case of suspicion of progressive disease, the hysterectomy will immediately take place. Peripheral blood and tumor samples will be used to explore dynamics of tumor and immune responses during therapy.

Follow-up: Adverse events will be followed up to 6 months after the final pembrolizumab administration. Outside the study protocol patients will be followed-up according SoC guidelines for uterine cancer. Patients will be asked to participate in follow-up of disease progression (2-year recurrence-free survival).

Study population: Primary MMRd UC patients at high-risk of recurrence (endometrioid grade 3 or clear cell histology) who are intended to be treated with a hysterectomy.

Intervention: Pembrolizumab, 200mg IV Q3W for a total of 9 administrations per patient, prior to SoC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed primary diagnosis of G3/CC MMRd uterine cancer who are intended to be treated with hysterectomy.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, is not a woman of childbearing potential (WOCBP) or agrees to follow contraceptive guidance during the treatment period and at least until standard-of-care hysterectomy.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

Exclusion Criteria:

* A WOCBP who has a positive serum pregnancy test at screening.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.
* Has received prior radiotherapy within 2 weeks of start of study treatment or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease with a 1-week washout is permitted.
* Has received a live vaccine or live-attenuated vaccine within 30 days before to the first dose of study intervention. Administration of killed vaccines and Covid vaccines is allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid).
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Establish fraction of patients that achieve major pathologic response | Tumor tissue is collected during standard of care hysterectomy (6 months after baseline)
  The primary objective of this phase 2 trial is to establish the fraction of patients that achieve a major pathologic response (MPR) after 9 cycles of pembrolizumab, with the ultimate aim of informing a follow-up randomized trial. MPR was chosen as primary endpoint to align with ongoing randomized phase 3 ICB trials on neo-adjuvant vs. adjuvant treatment in other tumor types (e.g. the NADINA trial in melanoma; NCT04949113).

SECONDARY OUTCOMES:
Radiologic response | MRI is scheduled before start study drug (week 4), during treatment (week 11, 17, and 23) and before surgery (week 32)
  To establish the objective response rate by radiologic assessment using MRI and RECIST1.1.
Recurrence Free Survival | RFS will be assessed 2 years after baseline
  To establish recurrence free survival (RFS) defined as the number of patients alive without any progress or recurrence at 2 years from disease diagnosis
Safety and tolerability (Adverse Events) | Through study completion, an average of 6 months per patient
  Adverse events will be documented according CTCAE

OTHER OUTCOMES:
The nature of the immune responses during treatment. | Will be determined after study completion, an average of 1 year
The involvement of TDLN in the immune responses on-treatment | Will be determined after study completion, an average of 1 year
Changes in circulating tumour DNA (ctDNA) during treatment | Will be determined after study completion, an average of 1 year
Pipelle biopsy as a predictor for response | Will be determined after study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans W Nijman, Prof. dr., Principal Investigator — University Medical Center Groningen, UMCG; Mathilde Jalving, Dr., Principal Investigator — University Medical Center Groningen, UMCG
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No